CLINICAL TRIAL: NCT02698514
Title: The Ratio of Hypnotic to Analgesic Potency of Sevoflurane and Desflurane : Randomized Controlled Trial
Brief Title: The Ratio of Hypnotic to Analgesic Potency of Volatile Anesthetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoungho Ryu, Clinical assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-12-023
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia was maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia was maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia was maintained with sevoflurane in patients undergoing standardized nociceptive stimulus (long-lasting tetanic stimulus of the ulnar nerve; 30 s, 50 mA, 50 Hz, square-wave).
  Other Names: SEVO
  Arms: Sevoflurane
Drug: Desflurane — Anesthesia was maintained with desflurane in patients undergoing standardized nociceptive stimulus (long-lasting tetanic stimulus of the ulnar nerve; 30 s, 50 mA, 50 Hz, square-wave).
  Other Names: DES
  Arms: Desflurane

SUMMARY:
The aim of this clinical trial is to evaluate the ratio of hypnotic to analgesic potency of sevoflurane and desflurane at equi-minimum alveolar concentration using SPI and EEG analysis.

DETAILED DESCRIPTION:
Anesthetic agents vary in their relative hypnotic potency. Recent studies demonstrated that equi-minimum alveolar concentration of various volatile anesthetic agents may produce different spectral entropy or bispectral index values. However, there is no study that demonstrate the difference between analgesic potency of volatile anesthetics. The aim of this clinical trial is to evaluate the ratio of hypnotic to analgesic potency of sevoflurane and desflurane at equi-minimum alveolar concentration using SPI and EEG analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia using volatile anesthetics and supraglottic airway (I-gel™)
* patients with american society of anesthesiologist physical status I, II
* patients aged 19-65 years
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients who had received any medication affecting the central nervous system
* patients who had received medication affecting the sympathetic or parasympathetic nervous systems
* patients undergoing tracheal intubation for airway management
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
Surgical pleth index | the 10 min at steady-state anesthesia after endotracheal intubation
  The analgesic potency of volatile anesthetics was evaluated by surgical pleth index during standardized nociceptive stimulus (30 s, 50 mA, 50 Hz tetanic stimulation).

SECONDARY OUTCOMES:
Bispectral index | the 10 min at steady-state anesthesia after endotracheal intubation
  The hypnotic potency of volatile anesthetics was evaluated by bispectral index during standardized nociceptive stimulus (30 s, 50 mA, 50 Hz tetanic stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea